CLINICAL TRIAL: NCT04135521
Title: Far Eastern Memorial Hospital
Brief Title: Dose-dense Chemotherapy Versus Intraperitoneal Chemotherapy as First-line Chemotherapy in Advanced Ovarian Cancer
Status: Completed | Type: Observational
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Sheng-Mou Hsiao, Chief of Department of Obstetrics & Gynecology, Associate Professor, Far Eastern Memorial Hospital
Other Study IDs: 108137-E
Record Dates: First submitted 2019-10-19; First posted 2019-10-22 (Actual); Last update posted 2020-06-29 (Actual); Status verified 2020-06

CONDITIONS: Advanced Ovarian Cancer
MeSH Terms: interventions — Hyperthermic Intraperitoneal Chemotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Intraperitoneal chemotherapy — Intraperitoneal or intravenous dose-dense platinum/taxane chemotherapy
  Other Names: Intravenous dose-dense chemotherapy

SUMMARY:
To compare dose-dense chemotherapy with intraperitoneal chemotherapy in patients with advanced stage ovarian cancer.

DETAILED DESCRIPTION:
Women aged 20 and above, diagnosed with advanced stage ovarian cancer (FIGO stage II~IV), who had received debulking surgery, followed by adjuvant chemotherapy (either dose-dense or intraperitoneal) at our institution between 01 January 2006 and 31 December 2018 were included in the study. Patient characteristics, any treatment related side-effects (peri-operative and post-operative complications, chemotherapy related adverse events), treatment response (complete or partial response, stable disease or progressive disease), post-treatment surveillance (disease status: disease-free, recurrence or cancer-related death) will be recorded. Univariate and multivariate logistic regression analysis will be employed to evaluate the survival benefit of the two different chemotherapy methods.

ELIGIBILITY:
Inclusion Criteria:

* Women with FIGO stage II~IV ovarian cancer
* At least one cycle of intravenous dose-dense or intraperitoneal chemotherapy had been administered as the front-line chemotherapy.

Exclusion Criteria:

* none

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — advanced ovarian cancer woman
Study Population: All consecutive women, who underwent intravenous dose-dense or intraperitoneal chemotherapy as the front-line chemotherapy were reviewed.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-10-28 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Progression-free survivals between this intraveous and intraperitoneal chemotherapy groups | 10 years
  months

SECONDARY OUTCOMES:
Overall survivals between this two groups | 10 years
  months

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Obstetrics and Gynecology, Far-Eastern Memorial Hospital, Banqiao District, New Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2019-10-22): https://cdn.clinicaltrials.gov/large-docs/21/NCT04135521/Prot_000.pdf